CLINICAL TRIAL: NCT04729036
Title: Interfragmentary Gap Discrepancy After Intraoral One-plate Fixation in Mandibular Angle Fracture
Brief Title: Mandibular Angle Fracture and Interframents Gap
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohsen, lecturer of oral and maxillofaciall surgery, Fayoum University
Other Study IDs: 29/12/2019
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Mandibular Fractures
MeSH Terms: conditions — Mandibular Fractures | interventions — Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mandibular fracture group
  Interventions: Procedure: open reduction and internal fixation

INTERVENTIONS:
Procedure: open reduction and internal fixation — The same surgical team have treated all the patients through open reduction via an intra-oral mucosal flap under general anesthesia with insertion and fixation of a 4-6 holes 2.0 miniplate and 5 mm screws at the superior border of the mandible at Champy's osteosynthesis line

SUMMARY:
Twenty-five patients with mandibular angle fracture were subjected to reduction and fixation through intra-oral open reduction and semi-rigid min plate fixation near the superior border of the mandible at Champy's osteosynthesis line. The linear inter-fragmentary gap was measured at the inferior border of the mandible after fixation of the fractured bony segments in the final aligned position immediately postoperative on a panoramic radiograph for the mesio-distal plane and a cone beam computed tomography for the bucco-lingual plane to assess any lingual splay. The healing process was clinically followed for 3 months postoperatively for any complications and/or patient complains

ELIGIBILITY:
Inclusion Criteria:

* minimally displaced mandibular angle fracture which needed intervention via reduction and fixation *medically free

Exclusion Criteria:

* - Patients with multiple mandibular fractures or patients with concomitant maxillary fracture.
* Patients with severely displaced mandibular angle fracture needing extra-oral open reduction and fixation.
* Medically compromised patients and patients with abnormalities that impair bone healing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: . All the patients suffered from minimally displaced mandibular angle fracture which needed intervention via reduction and fixation
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
interfragment gap | 3 months
  measure the mesio-distal plane discrepancy in terms of linear inter-fragmentary gap at the inferior border between the fractured mesial and proximal segments by CT

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University, Al Fayyum, Egypt